CLINICAL TRIAL: NCT00962897
Title: A Retrospective Review of Randomized Comparison of Prosthetic Femoropopliteal Bypass Versus Viabahn Endoprosthesis for Treatment of Symptomatic Femoral Artery Occlusion With Four Years Followup
Brief Title: Comparison of Prosthetic Femoropopliteal Bypass Versus Viabahn Endoprosthesis for Treatment of Symptomatic Femoral Artery Occlusion
Status: Completed | Type: Observational
Sponsor: Texas Vascular Associates (Other)
Collaborators: W.L.Gore & Associates (Industry)
Responsible Party: Dennis Gable, MD, Texas Vascular Associates/Baylor University Medical Center
Other Study IDs: 009-198, Viabahn #2
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Atherosclerosis; Lower Extremity Ischemia; Claudication; Rest Pain
Keywords: atherosclerosis; covered stent; percutaneous intervention; stent; angioplasty
MeSH Terms: conditions — Atherosclerosis; Intermittent Claudication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Surgical Bypass Group: Those patients that underwent bypass of blockage in the thigh with surgery.
  Interventions: Procedure: Femoral-popliteal bypass
- Stent-graft group: Patients that underwent treatment of blockage in the thigh with balloon angioplasty and stent placement.
  Interventions: Procedure: Stent-graft placement

INTERVENTIONS:
Procedure: Femoral-popliteal bypass — Surgical bypass of blockage in the thigh
  Groups: Surgical Bypass Group
Procedure: Stent-graft placement — Patients that underwent treatment of blockage in the thigh arteries with balloon angioplasty with stent-graft placement.
  Groups: Stent-graft group

SUMMARY:
A retrospective review with four year followup on patients that had previously been enrolled in a study to evaluate blockages in the lower legs. The study looked at patients that had undergone a bypass of the leg from the groin to the knee area with an incision in each area using general anesthesia. These patients were compared to others who had undergone treatment with balloon dilatation and stents in the arteries in the thighs with only numbing medicine. The study was completed two years ago and was initially designed to look at outcomes at 24 months. Now the investigators are trying to go back and look at outcomes of these patients' treatment at 4 years by simply reviewing their records.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic lower extremity ischemia patients treated by femoral-popliteal bypass or percutaneous covered stent graft in previous prospective study

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vascular surgery clinic patients with ischemic symtpom of the lower extremities. Patients were previously enrolled in a randomized prospective study comparing treatment of blockage in the legs with a surgical bypass or percutaneous covered stent placemnt.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2003-09; Primary Completion 2007-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Primary artery/graft patency | 48 months

SECONDARY OUTCOMES:
Secondary artery/graft patency | 48 months
Limb salvage | 48 months
Improvement of lower extremity ischemic symptoms | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Dennis R Gable, M.D., Principal Investigator — Texas Vascular Associates
Locations (1):
- Texas Vascular Associates, Dallas, Texas, United States

REFERENCES:
- [Background] Alimi YS, Hakam Z, Hartung O, Boufi M, Barthelemy P, Aissi K, Dubuc M. Efficacy of Viabahn in the treatment of severe superficial femoral artery lesions: which factors influence long-term patency? Eur J Vasc Endovasc Surg. 2008 Mar;35(3):346-52. doi: 10.1016/j.ejvs.2007.09.005. Epub 2007 Nov 5. PMID 17983772
- [Background] Fischer M, Schwabe C, Schulte KL. Value of the hemobahn/viabahn endoprosthesis in the treatment of long chronic lesions of the superficial femoral artery: 6 years of experience. J Endovasc Ther. 2006 Jun;13(3):281-90. doi: 10.1583/05-1799.1. PMID 16784314
- [Result] McQuade K, Gable D, Hohman S, Pearl G, Theune B. Randomized comparison of ePTFE/nitinol self-expanding stent graft vs prosthetic femoral-popliteal bypass in the treatment of superficial femoral artery occlusive disease. J Vasc Surg. 2009 Jan;49(1):109-15, 116.e1-9; discussion 116. doi: 10.1016/j.jvs.2008.08.041. Epub 2008 Nov 22. PMID 19028055
- [Result] Kedora J, Hohmann S, Garrett W, Munschaur C, Theune B, Gable D. Randomized comparison of percutaneous Viabahn stent grafts vs prosthetic femoral-popliteal bypass in the treatment of superficial femoral arterial occlusive disease. J Vasc Surg. 2007 Jan;45(1):10-6; discussion 16. doi: 10.1016/j.jvs.2006.08.074. Epub 2006 Nov 28. PMID 17126520